CLINICAL TRIAL: NCT05150145
Title: A Prospective Phase II Randomized Clinical Study of Radiotherapy or Observation of Liver Metastases for Small Cell Lung Cancer.
Brief Title: Radiotherapy or Observation of Liver Metastases in Small Cell Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guizhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-SCLC-liver001
Record Dates: First submitted 2021-11-28; First posted 2021-12-08 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Radiotherapy; Complications
Keywords: Radiotherapy;liver metastases;Small cell lung cancer;

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiotherpy will be performed to thoracic and liver metastasis. (Experimental): Radiotherapy for liver metastases and thoracic will be performed in paticipants with liver metastasis who achieved CR or PR after chemotherapy.
  Interventions: Radiation: Radiotherpy will be performed to thoracic and liver metastasis after chemotherapy.
- Radiotherpy will be performed to thoracic. (No Intervention): Radiotherapy performed only on the thoracic after chemotherapy of paticipants with liver metastasis who achieved CR or PR.

INTERVENTIONS:
Radiation: Radiotherpy will be performed to thoracic and liver metastasis after chemotherapy. — Intensity modulated radiotherapy will be performed to liver metastasis and thoracic SCLC patients who achieved CR or PR after chemotherapy .
  Arms: Radiotherpy will be performed to thoracic and liver metastasis.

SUMMARY:
The aim of this randomized study is to investigate local tumor control,survival outcomes and complications on patients of liver metastasis in small cell lung cancer.

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) is a kind of disease with high degree of malignancy and poor prognosis.Based on the effectiveness of systemic chemotherapy, the treatment of primary lesions and whole brain radiotherapy can bring survival benefits to patients with extensive stage small cell lung cancer.Patients with liver metastasis have a worse prognosis than those with other organ metastases.Local radiotherapy for patients with liver metastasis may have a better prognosis.However, clinical data of the safety and efficacy of whole liver radiotherapy for liver metastasis are still lacking.The purpose of this prospective study is to evaluate the safety, efficacy, and tolerability of liver metastatic radiotherapy in small cell lung cancer (SCLC).

ELIGIBILITY:
Inclusion Criteria

1. Informed consent (radiation, medication) before treatment;
2. Age 18 to 70 years old,regardless of gender;
3. Initial SCLC confirmed by histopathological or cytological examination;
4. Metastatic lesions in the distant area: included liver metastasis；
5. Physical status score ECOG: 0 to 2；
6. The expected survival time is more than 3 months;
7. Bone marrow function:hemoglobin(HGB)>90g/L,platelet(PLT)>100×109/L,neutrophil cell(WBC)>1.5×109/L(*normal value);
8. Liver function:alanine aminotransferase(ALT) and aspertate aminotransferase(AST)<1.5 times of the upper limit of normal(ULN);Total bilirubin <1.5ULN;
9. Renal function:Serum creatinine was lower than 1.5ULN,and the endogenous creatinine clearance rate(Ccr) is higher than 55mL/min;
10. Initial treatment (previously did not receive any thoracic radiotherapy or surgery).

Exclusion Criteria:

1. patients with history of mental illness;
2. patients combined with other malignancies;
3. Active period of disease caused by bacteria, fungi or viruses; and these severe infection requiring intravenous antibiotics,antifungal or antiviral therapy;
4. Patients with serious cardiovascular disease ,including uncontrolled hypertension, unstable angina,history of myocardial infarction within the past 12 months,and severe arrhythmias.
5. Patients with poorly controlled diabetes who are judged to be unfit for chemotherapy by doctors.
6. History of hepatitis and cirrhosisi ;
7. pregnant, lactating patients;
8. Patients with poor compliance；
9. Researchers believe that it is not appropriate to participate in this test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Intrahepatic progression -free survial(Intrahepatic-PFS) | UP to 5years
  Intrahepatic progression -free survial is defined as the duration of time from start of treatment to time of progression of hepatic metastasis.
Overall survival (OS) | UP to 5years
  Overall survival is defined as the time interval from date of diagnosis to date of death from any cause.

SECONDARY OUTCOMES:
Progression-free survival(PFS) | UP to 5years
  PFS is defined as the duration of time from start of treatment to time of progression or death,whichever occurs first.
Adverse events(toxicities) | UP to 5years
  The descriptions and grading scales found in the revised Common Terminology Criteria for Adverse Events(CTCAE 4.0) will be utilized for all toxicity reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Shengfa Su, doctor, Principal Investigator — Affiliated Hospital of Guizhou Medical University
Locations (1):
- The affiliated hospital of Guizhou medical university, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: No